CLINICAL TRIAL: NCT06775990
Title: The Evaluation of Current Molecules and Receptor Profiles Associated with Pediatric Obesity
Brief Title: Molecules Associated with Pediatric Obesity
Acronym: Thesis
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Scientific Research Project Coordination Unit of Istanbul University-Cerrahpasa (Unknown)
Responsible Party: Principal Investigator, Ezgi Kürkçü Kahraman, Assistant Prof., Istanbul University - Cerrahpasa
Other Study IDs: 34574; 34574 (Other Grant/Funding Number: Istanbul University-Cerrahpasa)
Record Dates: First submitted 2025-01-04; First posted 2025-01-15 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: OBESITY
Keywords: Child; Obesity; Obesity parameters and receptors
MeSH Terms: conditions — Obesity | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples With DNA — Serum samples were stored at -80 degrees Celsius.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy control: Children between the ages of 06-18 years without acute or chronic diseases and without major congenital anomalies were included in the study. Two groups were formed from 30 obese children with BMI values above the 95th percentile according to the WHO criteria accepted by the Ministry of Health and 60 healthy children with BMI values between the 85th and 15th percentiles who constituted the control group. Of the 60 children, 35 were girls and 25 were boys.
  Serum leptin, leptin receptor (LEPR), ghrelin, acylated ghrelin, deacylated ghrelin, ghrelin receptor (GHSR), kisspeptin (KISS1), kisspeptin receptor (KISS1R), preptin, Peroxisome proliferator-activated receptor gamma (PPAR γ), nod-like receptor pyrin domain-containing 3 (NLRP3), interleukin-18 (IL-18) levels were determined by ELISA in thirty obese and thirty healthy children.
  Interventions: Other: Blood sample
- Obese children.: Children between the ages of 06-18 years without acute or chronic diseases and without major congenital anomalies were included in the study. Two groups were formed from 30 obese children with BMI values above the 95th percentile according to the WHO criteria accepted by the Ministry of Health and 60 healthy children with BMI values between the 85th and 15th percentiles who constituted the control group. Of the 60 children, 35 were girls and 25 were boys. Serum leptin, leptin receptor (LEPR), ghrelin, acylated ghrelin, deacylated ghrelin, ghrelin receptor (GHSR), kisspeptin (KISS1), kisspeptin receptor (KISS1R), preptin, Peroxisome proliferator-activated receptor gamma (PPAR γ), nod-like receptor pyrin domain-containing 3 (NLRP3), interleukin-18 (IL-18) levels were determined by ELISA in thirty obese and thirty healthy children.
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Children were not given any medication in the study. Peripheral blood samples from the children were collected, centrifuged and stored in the biochemistry laboratory in deep freezers at -80 degree celcius. From stored serum samples leptin, leptin receptor (LEPR), ghrelin, acylated ghrelin, deacylated ghrelin, ghrelin receptor (GHSR), kisspeptin (KISS1), kisspeptin receptor (KISS1R), preptin, Peroxisome proliferator-activated receptor gamma (PPAR γ), nod-like receptor pyrin domain-containing 3 (NLRP3), interleukin-18 (IL-18) levels were determined by ELISA in thirty obese and thirty healthy children.

SUMMARY:
Childhood obesity is linked to obesity in adulthood and causes severe problems, particularly due to its relationship with metabolic syndrome, diabetes, cancer, and cardiovascular diseases. The determination of markers and receptor profiles related to parameters contributing to energy homeostasis in healthy children with a normal body mass index and children with obesity will guide the diagnosis and treatment of pediatric obesity. The aim was to determine possible relationships by evaluating markers contributing to energy homeostasis in healthy individuals and children with obesity.

Anthropometric measurements of the children were obtained. The serum leptin, leptin receptor (LEPR), ghrelin, acylated ghrelin, deacylated ghrelin, ghrelin receptor (GHSR), kisspeptin (KISS1), kisspeptin receptor (KISS1R), preptin, peroxisome proliferator activated receptor gamma (PPARγ), nod-like receptor pyrin domain-containing 3 (NLRP3), and interleukin-18 (IL-18) levels of thirty children with obesity and thirty healthy children were determined using ELISA.

DETAILED DESCRIPTION:
Children between the ages of 6 and 18 years without acute or chronic diseases and without major congenital anomalies were included in the study. Peripheral blood samples were collected from children admitted to Tekirdağ Namık Kemal University Faculty of Medicine, Department of Pediatrics after 8-12 hours of fasting. Two groups were formed from 30 children with obesity BMI values above the 95th percentile according to the WHO criteria accepted by the Ministry of Health and 30 children with healthy BMI values between the 85th and 15th percentiles who constituted the control group. Of the 60 children, 35 were girls and 25 were boys.

Before the study, Ethics Committee approval documents numbered 2020.01.01.01 were obtained from Tekirdağ Namık Kemal University where the study was conducted. The families of the children, especially their parents, were informed. After a detailed pediatric physical examination and informing them about their inclusion in the study, signed consent forms from the consenting parents were obtained, and the children were informed verbally. Peripheral blood samples obtained from the children were collected, centrifuged, and stored in the biochemistry laboratory in deep freezers at -80°C.

The weights, heights, and waist, hip, head, and neck circumferences (Cs) of all the children were measured and recorded. BMI, waist/hip ratios, and other ratios and formulas related to obesity were calculated from anthropometric measurements, and statistical analyses of the anthropometric measurements of controls and children with obesity were performed.

NLRP3, leptin, acylated ghrelin, deacyl ghrelin, preptin, PPAR γ, LEPR, GHSR, KISS1R, and IL-18 were analyzed by the sandwich ELISA method, and ghrelin and KISS1 parameters were analyzed by the competitive ELISA method in the control and obese groups.

In the statistical evaluation of the data, parametric or nonparametric statistical tests appropriate for the distribution characteristics of the data obtained were applied. The Shapiro-Wilk test was used to determine whether the values of the parameters conformed to a normal distribution. Independent samples t tests, Mann-Whitney U tests, and Kruskal-Wallis tests were used to evaluate the differences between the groups, and Pearson and Spearman correlation analyses were performed to examine whether the values of the parameters changed together. In addition, the Mann-Whitney U test was applied with the Bonferroni correction in the evaluation of subgroups.

Statistical analyses were performed with SPSS (Statistical Package for the Social Sciences) Version 26. The means, standard deviations, standard errors, and medians were compared between the control and obese groups. The statistically significant difference between them was evaluated according to whether the values showed a parametric or nonparametric distribution. P values less than 0.05 were considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-18 years were included in the study
* 30 obese children with BMI values above the 95th percentile according to WHO criteria and 30 healthy children with BMI values between the 85th and 15th percentiles and 60 healthy children with anorexia were included in the study
* Children without acute or chronic diseases and without major congenital anomalies were included in the study.

Exclusion Criteria:

* Be over 18 years of age
* Presence of conditions that may cause secondary obesity, such as hypothyroidism or polycystic ovary syndrome
* Children with previous bariatric surgery or repeated diet attempts;
* Children with a serious acute or chronic illness (active infection, heart failure, cardiovascular disease, cerebrovascular disease, acute renal failure, chronic renal failure, chronic lung disease, malignancy) were excluded.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children between the ages of 6 and 18 years without acute or chronic diseases and without major congenital anomalies were included in the study. Peripheral blood samples were collected from children admitted to Tekirdağ Namık Kemal University Faculty of Medicine, Department of Pediatrics after 8-12 hours of fasting. Two groups were formed from 30 children with obesity BMI values above the 95th percentile according to the WHO criteria accepted by the Ministry of Health and 30 children with healthy BMI values between the 85th and 15th percentiles who constituted the control group. Of the 60 children, 35 were girls and 25 were boys.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Obesity BMI values according to WHO criteria accepted by the Ministry of Health | 6 months
  Two groups were formed from 30 children with obesity BMI values above the 95th percentile according to the WHO criteria accepted by the Ministry of Health and 30 children with healthy BMI values between the 85th and 15th percentiles who constituted the control group.
  Weight in kilograms Height in meters weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi Kürkçü Kahraman, Assist Prof., Principal Investigator — Istanbul Beykent University
Locations (1):
- Namik Kemal University, Tekirdağ, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Case Reports Metabolism . 2021 Mar:116:154438. doi: 10.1016/j.metabol.2020.154438. Epub 2020 Nov 19. — https://pubmed.ncbi.nlm.nih.gov/33221380/